CLINICAL TRIAL: NCT01795014
Title: Analysis of the Relationship Between Optic Nerve Sheath Diameter and the Spontaneous Venous Pulsation in Primary Open-angle Glaucoma
Brief Title: Correlation of Orbital Cerebrospinal Fluid Pressure and Retinal Venous Outflow in Primary Open-angle Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: SVP0002
Record Dates: First submitted 2013-02-12; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Primary Open Angle Glaucoma; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls: Healthy volunteers with no family history of glaucoma, an increased or asymmetrical cup/disc ratio or any other optic disc structural change (notching, disc hemorrhage) or an IOP above 21 mmHg that could suggest possible glaucoma suspects.
- Primary open-angle Glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at least one measurement of IOP of >21 mmHg required
- Normal Tension Glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at maximum recorded IOP of < 21 mmHg

SUMMARY:
A spontaneous venous pulsation over the optic disc is an ophthalmological sign that can potentially be found in up to 98% of healthy individuals. In fact, the lack of this spontaneous retinal venous pulse has been consistently implicated as an indicator of a more advanced form of certain ocular diseases, specifically open-angle glaucoma. However, the mechanisms behind these change in the retinal venous system are not clear. Some evidence suggests that extraocular features such as intracranial pressure (ICP) may play a role in regulating the intraocular venous outflow. The reasons for this hypothetical downstream resistance to venous outflow are not fully understood, with advances in this field being limited by our technological-imposed difficulties in assessing the structures behind the globe.

However, it has been established that the volume of cerebrospinal fluid surrounding the optic nerve correlates with the ICP at the orbital level. Recent studies have suggested that non-invasive ultrasound-based recordings have correlated this surrogate for orbital ICP with the intraocular pressure (IOP) in glaucoma patients with an otherwise normal IOP range (normal tension glaucoma - NTG).

The investigators will therefore conduct a test to determine if this cerebrospinal volume surrounding the optic nerve correlates with the frequency of observation of an otherwise signal of venous dysfunction (i.e. the lack of a visible pulse in the retinal central vein) Additionally, the investigators will assess if this correlation is different between healthy individuals, hypertensive primary-open angle glaucoma or NTG patients.

DETAILED DESCRIPTION:
1. Spontaneous venous pulsation will be recorded after a one minute fundoscopy observation.
2. B-mode ultrasound of the orbit will be performed and the optic nerve sheath diameter measured 3mm behind the globe
3. Visual field examination will be performed.
4. Structural examination of the optic disc (confocal microscopy) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply with the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for cataract surgery)
* eye disease (except glaucoma)
* systemic diseases with ocular involvement like diabetes or graves ophthalmopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Spontaneous venous pulsation | Up to 3 months
  Assessing whether the frequency of the spontaneous venous pulsation phenomenon is associated with the optic nerve sheath diameter in glaucoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- KU Leuven, Leuven, Flemish Brabant, Belgium